CLINICAL TRIAL: NCT00149682
Title: Obesity Assessment and Education Through the Internet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: OAEI (completed)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: 6-month educational program
Behavioral: 6-month standard care program

SUMMARY:
The purpose of this study is to develop a web-based obesity risk assessment and counseling tool and examine its feasibility and effectiveness in improving the rate and quality of physician counseling about obesity, dietary change, and physical activity.

DETAILED DESCRIPTION:
Despite the high prevalence of obesity and its associated health risks, physicians do not address weight and behaviors that contribute to obesity because of lack of knowledge, training, and access to resources. To address these physician barriers to counseling, the investigator has developed a web-based tool that collects and integrates relevant patient clinical and behavioral information online and generates patient-specific recommendations and links to resources in the form of electronic patient and physician reports. In doing so, the tool provides physicians with a time saving device that identifies at risk patients who are motivated to make behavioral changes; at the same time, the tool provides tailored resources and recommendations that help physicians deliver more effective counseling.

The pilot study described in this application randomizes overweight primary care patients to a control group and the web-based intervention. The aims of the study are to examine the feasibility of incorporating the web-based tool into primary care practice and to collect preliminary data on its potential effectiveness on improving the rate and quality of physician-patient discussions about weight and on improving several clinical and behavioral outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Received invitation from participating primary care practices
* Scheduled non-urgent appointment with their usual primary care provider
* BMI > 25 kg/m2
* Willing and able to participate in a web-based computerized self-administered questionnaire
* English-speaking

Exclusion Criteria:

* Pregnancy
* Terminal illness
* Not competent to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-07; Study Completion 2007-12

PRIMARY OUTCOMES:
Physician counseling about weight and weight-related behaviors

SECONDARY OUTCOMES:
Changes in cardiovascular risk factors
Improvements in physical activity and dietary behavior

CONTACTS AND LOCATIONS:
Overall Officials: Christina C. Wee, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Wee CC, Davis RB, Phillips RS. Stage of readiness to control weight and adopt weight control behaviors in primary care. J Gen Intern Med. 2005 May;20(5):410-5. doi: 10.1111/j.1525-1497.2005.0074.x. PMID 15963162